CLINICAL TRIAL: NCT03662685
Title: Immunogenetic Profiling of Goeckerman Therapy in the Treatment of Psoriasis Vulgaris
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closing of the Goeckerman program at UCSF and loss of funding, PI left UCSF
Sponsor: University of California, San Francisco (Other)
Collaborators: National Psoriasis Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Goeckerman Immunogenetics
Record Dates: First submitted 2017-10-05; First posted 2018-09-07 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Psoriasis Vulgaris; Psoriasis
Keywords: goeckerman; phototherapy; psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Phototherapy; Coal Tar

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Goeckerman Therapy (Active Comparator): Patients with psoriasis who will receive Goeckerman therapy 5 days per week for 6 weeks.
  Interventions: Other: Goeckerman Therapy
- Phototherapy Only (Active Comparator): Patients with psoriasis who will receive narrowband ultraviolet B (NB-UVB) phototherapy 3 days per week for 12 weeks.
  Interventions: Device: Phototherapy Only
- Crude Coal Tar Only (Active Comparator): Patients with psoriasis who will receive skin treatment with crude coal tar only 5 days per week for 6 weeks.
  Interventions: Drug: Crude Coal Tar Only

INTERVENTIONS:
Other: Goeckerman Therapy — The Goeckerman regimen consists of exposure to narrowband ultraviolet B (NB-UVB) light phototherapy and application of crude coal tar to the skin 5 days per week. The treatment will occur the UCSF outpatient skin treatment center for approximately 4-5 hours, 5 days a week for 6 weeks (total of 30 sessions). The treatment is consistent with the standard of care Goeckerman treatment protocol at UCSF.
  Other Names: Combination Treatment with Phototherapy and Crude Coal Tar; Goeckerman Regimen
  Arms: Goeckerman Therapy
Drug: Crude Coal Tar Only — A topical medication consisting of crude coal tar will be applied to the psoriatic skin under plastic wrap occlusion for approximately up to 4-5 hours, 5 days a week for 6 weeks (total of 30 sessions), at the outpatient skin treatment center at UCSF.
  Other Names: Coal tar
  Arms: Crude Coal Tar Only
Device: Phototherapy Only — Light treatment with narrowband ultraviolet B (NB-UVB) phototherapy three days per week for 12 weeks at the UCSF Phototherapy Center per the standard UCSF phototherapy protocol, in which starting dose is based on the subject's Fitzpatrick skin type and gradually increased as tolerated. Each phototherapy treatment will last approximately from under 1 minute to less than 15 minutes.
  Other Names: Ultraviolet B; Narrowband ultraviolet B; NB-UVB; UVB phototherapy; Phototherapy; Light treatment
  Arms: Phototherapy Only

SUMMARY:
This study examines the effect of Goeckerman therapy (a combination of phototherapy and topical crude coal tar), crude coal tar alone, and phototherapy alone on the immunologic and genetic environment within psoriatic skin lesions.

DETAILED DESCRIPTION:
This is a three-arm, open-label study to examine the effect of Goeckerman therapy. Goeckerman therapy is known for its high efficacy and favorable safety profile in the treatment of psoriasis. It consists of a combination of phototherapy and topical crude coal tar). This study will examine how Goeckerman therapy, crude coal tar alone, and phototherapy alone affect the mmunologic and genetic environment within psoriatic skin lesions. Fifteen subjects with moderate to severe psoriasis will be enrolled. Biopsy samples will be collected and undergo molecular profiling to further elucidate the mechanism of action by which Goeckerman treatment improves psoriatic skin lesions.

ELIGIBILITY:
Inclusion criteria

1. Male or female ≥ 18 years of age at enrollment.
2. Documentation of predominately moderate to severe plaque psoriasis for at least 6 months prior to enrollment.
3. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
4. Subject is considered a candidate for phototherapy or systemic therapy
5. Body Surface Area (BSA) ≥ 5%.
6. Physical exam within clinically acceptable limits.

Exclusion criteria

1. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
2. Subject has predominantly non-plaque form of psoriasis.
3. Subject has drug-induced psoriasis.
4. Subject with current, or a history of, severe psoriatic arthritis well controlled on current therapy.
5. Patient has absolute or relative contraindication to phototherapy, including photosensitizing disorders.
6. Evidence of abnormality of any immune cell population from a drug-induced or genetic cause.
7. Known HIV positive status.
8. Known allergy to lidocaine, other local anesthetics, or any component of local anesthetic agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Number of differentially expressed immune cell populations | 12 weeks
  Perform quantitative analysis of the immunologic and genetic changes in immune cell populations after treatment with traditional Goeckerman (NBUVB + coal tar), coal tar only, and NB-UVB only, at weeks 2, 4, and 12 compared to baseline week 0. The immunologic profiles will be compared between subjects receiving the traditional Goeckerman therapy (NB-UVB + coal tar), coal tar only, and NB-UVB therapy only.

SECONDARY OUTCOMES:
Number of differentially expressed genes and pathways | 12 weeks
  Quantify the number of differentially expressed genes in each cell population by RNA-sequencing at weeks 0, 2, 4, 12 after receiving traditional Goeckerman therapy (NB-UVB + coal tar), coal tar only, and NB-UVB therapy only.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Bhutani, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Psoriasis and Skin Treatment Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta R, Debbaneh M, Butler D, Huynh M, Levin E, Leon A, Koo J, Liao W. The Goeckerman regimen for the treatment of moderate to severe psoriasis. J Vis Exp. 2013 Jul 11;(77):e50509. doi: 10.3791/50509. PMID 23892536
- [Background] Menter A, Cram DL. The Goeckerman regimen in two psoriasis day care centers. J Am Acad Dermatol. 1983 Jul;9(1):59-65. doi: 10.1016/s0190-9622(83)70107-6. PMID 6886105
- [Background] Moscaliuc ML, Heller MM, Lee ES, Koo J. Goeckerman therapy: a very effective, yet often forgotten treatment for severe generalized psoriasis. J Dermatolog Treat. 2013 Feb;24(1):34-7. doi: 10.3109/09546634.2012.658014. Epub 2012 Mar 4. PMID 22329632
- [Background] van den Bogaard EH, Bergboer JG, Vonk-Bergers M, van Vlijmen-Willems IM, Hato SV, van der Valk PG, Schroder JM, Joosten I, Zeeuwen PL, Schalkwijk J. Coal tar induces AHR-dependent skin barrier repair in atopic dermatitis. J Clin Invest. 2013 Feb;123(2):917-27. doi: 10.1172/JCI65642. Epub 2013 Jan 25. PMID 23348739
- [Background] Li B, Tsoi LC, Swindell WR, Gudjonsson JE, Tejasvi T, Johnston A, Ding J, Stuart PE, Xing X, Kochkodan JJ, Voorhees JJ, Kang HM, Nair RP, Abecasis GR, Elder JT. Transcriptome analysis of psoriasis in a large case-control sample: RNA-seq provides insights into disease mechanisms. J Invest Dermatol. 2014 Jul;134(7):1828-1838. doi: 10.1038/jid.2014.28. Epub 2014 Jan 17. PMID 24441097
- [Background] Gupta R, Ahn R, Lai K, Mullins E, Debbaneh M, Dimon M, Arron S, Liao W. Landscape of Long Noncoding RNAs in Psoriatic and Healthy Skin. J Invest Dermatol. 2016 Mar;136(3):603-609. doi: 10.1016/j.jid.2015.12.009. Epub 2015 Dec 18. PMID 27015450
- [Background] Sekhon S, Jeon C, Nakamura M, Afifi L, Yan D, Wu JJ, Liao W, Bhutani T. Review of the mechanism of action of coal tar in psoriasis. J Dermatolog Treat. 2018 May;29(3):230-232. doi: 10.1080/09546634.2017.1369494. Epub 2017 Sep 19. PMID 28814117
- [Background] Zhu TH, Nakamura M, Farahnik B, Abrouk M, Singh RK, Lee KM, Hulse S, Koo J, Bhutani T, Liao W. The Patient's Guide to Psoriasis Treatment. Part 4: Goeckerman Therapy. Dermatol Ther (Heidelb). 2016 Sep;6(3):333-9. doi: 10.1007/s13555-016-0132-7. Epub 2016 Jul 29. PMID 27474032